CLINICAL TRIAL: NCT04450927
Title: Data Collection of Standard Care and Evaluation of NHLBI Patients and Donors
Status: Enrolling by invitation | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 200099; 20-H-0099
Record Dates: First submitted 2020-06-27; First posted 2020-06-30 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12-03

CONDITIONS: Wide Spectrum of Diseases; Hematologic Diseases
Keywords: Repository; Hematology; Cardiology; Pulmonary; Oncology; Natural History
MeSH Terms: conditions — Hematologic Diseases; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Data collection and treatment according to guidelines of standard of medical evaluation and care. No investigational treatments or procedures will be administered on this protocol.

SUMMARY:
Background:

Researchers seek ways to study people s medical problems in order to teach and further general knowledge. The ability to assess and treat people with a wide range of diseases is critical to training people to be good doctors. It is also needed to keep medical staff up to date. In this study, researchers want to study the course of some illnesses to learn more about them. To do this, they will collect and review people s medical records. In some cases, they may also provide treatment.

Objective:

To collect data that may be used to help researchers create ideas for future research.

Eligibility:

People age 2 and older who have or are suspected to have a medical condition for which they have been referred to NIH s National Heart, Lung, and Blood Institute, as well as stem cell donors

Design:

Participants may be screened with a review of the following:

Medical records

Scans and images

Other existing samples and reports.

Participants medical data will be collected from the standard care they receive. This includes their routine blood and urine tests, X-rays and scans, and other tests to diagnose or follow their medical condition. Data will also be collected from the treatments they may receive. For stem cell donors, data from apheresis procedures will be collected. Demographic data will also be collected.

All of the data will be kept in the medical records or on secure network drives.

Some participants may need to be treated for their medical condition. If so, they will sign a separate consent form for that treatment.

Participation lasts up to 2 years.

DETAILED DESCRIPTION:
This protocol is designed to provide a repository of information to allow for hypothesis generation in future research. This information will be drawn from standard medical care/procedures and follow up of patients and healthy volunteers, including transplant donors, who are not currently receiving therapy on an active NHLBI research protocol. It allows investigation into the problems of these patients for the purpose of teaching and furthering general knowledge. The ability to evaluate and treat patients with a wide variety of diseases is critical to maintaining our accreditation with the hematology-oncology, cardiology, and pulmonary fellowship programs and training our fellows to be competent physicians, as well as for keeping all staff, including senior staff, up-to-date and familiar with the evaluation and treatment of patients with a wide spectrum of diseases. Periodic follow-up and treatment of patients previously entered on NHLBI protocols in order to monitor the long-term course of the underlying disease and the consequences of experimental treatments is also required for fellowship training, and for maintenance of good referral relationships with patients and their physicians. This study also allows for standard apheresis procedures for transplant donors and for care of volunteers who may present with a treatable condition.

ELIGIBILITY:
* ELIGIBILITY:

  1. Patients (including those referred to us to rule out a disease or condition) and stem cell donors, may be entered on this protocol at the discretion of the Principal and/or Associate Investigators.
  2. The patient or the patient's Legally Authorized Representative is capable of informed consent and signs the consent form. The consent form will be signed by parents or guardians of patients under the age of 18.
  3. Age more than or equal to 2 and weight > 12 kg

Ages: 2 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All subjects 2 or older and weighing greater than 12 kg, who meet inclusion criteria will be considered for participation on this protocol at this discretion of the Principal or Associate Investigator
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2020-06-16 (Actual); Primary Completion 2040-12-31 (Estimated); Study Completion 2040-12-31 (Estimated)

PRIMARY OUTCOMES:
To provide a repository of information on enrolled participants to allow for hypothesis generation in future research | 20 years
  To provide a repository of information on enrolled participants to allow for hypothesis generation in future research

SECONDARY OUTCOMES:
To add value to the NHLBI training program | 20 years
  To add value to the NHLBI training program by providing consult, treatment, diagnostic tests, and medical follow-up of participants

CONTACTS AND LOCATIONS:
Overall Officials: Georg Aue, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2020-H-0099.html